CLINICAL TRIAL: NCT04694820
Title: txt4TKI: An Innovative Mobile Intervention to Improve Tyrosine Kinase Inhibitor Management Among Chronic Myeloid Leukemia Patients
Brief Title: A Mobile Intervention (txt4TKI) for the Improvement of Tyrosine Kinase Inhibitor Management in Patients With Chronic Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20P.140; JT 14933 (Other: JeffTrial Number)
Record Dates: First submitted 2020-12-07; First posted 2021-01-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text message intervention (Experimental): Six month text message intervention
  Interventions: Other: Text Message-Based Navigation Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Text Message-Based Navigation Intervention — Receive txt4TKI
  Other Names: Automated Text Message-Based Navigation, Text Message-Based Navigation
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies the feasibility and acceptability of a mobile intervention called txt4TKI for the improvement of tyrosine kinase inhibitor management in patients with chronic myeloid leukemia. Tyrosine kinase inhibitors (TKI) are associated with numerous potential side effects, including a decrease in bone marrow activity (myelosuppression), nausea, diarrhea, fatigue, and soft-tissue swelling (edema), especially in the face and lower legs, which are the primary reasons for patients to discontinue TKI medication. Using a mobile text messaging (TXT) intervention that emphasizes the importance of TKI compliance may improve TKI adherence in patients with chronic myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* PHASE 1: Patients diagnosed with chronic myeloid leukemia
* PHASE 1: Initiated tyrosine kinase inhibitors therapy for a year
* PHASE 1: Able to read and understand English
* PHASE 1: Able to provide informed consent
* PHASE 1: Have a mobile phone with TXT capability
* PHASE 1: Know how to use TXT
* PHASE 2: Patients diagnosed with chronic myeloid leukemia in the chronic phase
* PHASE 2: Starting tyrosine kinase inhibitors therapy or has been on tyrosine kinase inhibitors with anticipation of at least 6 month duration of use
* PHASE 2: Able to read and understand English
* PHASE 2: Able to provide informed consent
* PHASE 2: Have a mobile device with TXT capability
* PHASE 2: Willing to use a wireless pill bottle during study for 6 months
* PHASE 2: Know or willing to learn how to use TXT

Exclusion Criteria:

• Cognitive impaired document in the electronic medical record (EMR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Assessment of TKI Treatment Date | Up to 6 months post-baseline
  Will be extracted from the electronic medical record (EMR) chart, including tyrosine kinase inhibitor (TKI) treatment initiation dates
Assessment of TKI Treatment change | Up to 6 months post-baseline
  Will be extracted from the electronic medical record (EMR) chart, including change of treatment.
Assessment of TKI Discontinuation | Up to 6 months post-baseline
  Will be extracted from the electronic medical record (EMR) chart, including discontinuing treatment
Feasibility of Compliance | Up to 6 months post-baseline
  Will be measured through study accrual, attrition, adverse event monitoring data, and system usage frequencies. 90% of the study participants adequately use the smart pill bottles will be acceptable. The intervention will be considered feasible if attrition does not exceed 30%. 90% of participant texting back to the system at least once will be considered adequate.
Acceptability of Mobile Involvement | Up to 6 months post-baseline
  Will be measured through a satisfaction measure and patient interview data. Acceptability will be established by a group median score >= 3 on the 1-4 satisfaction scale. Further, transcripts of the audio recorded post-intervention patient interviews will be analyzed using grounded theory and constant comparative methods. Analysis will examine patient perceptions of the usefulness and satisfaction with the txt4TKI intervention. After the research team reaches a consensus on a coding scheme, the principal investigator (PI) and the project manager will code independently the transcripts, examining patient's satisfaction with and evaluation of the txt4TKI intervention.
TKI adherence | Up to 6 months post-baseline
  Will be assessed by AdhereTech wireless smart pill bottes for all participants, which are Health Insurance Portability and Accountability Act (HIPAA)-compliant Food and Drug Administration (FDA) class I medical devices that monitor electronic tracking of bottle and percent of pills detected inside the bottle.
Symptom burden | Up to 6 months post-baseline
  The MD Anderson Symptom Inventory-Chronic Myeloid Leukemia (MDASI-CML) will be used to assess patient symptom burden.
Knowledge and self-efficacy for taking medication | Up to 6 months post-baseline
  Will be measured by the Medication Understanding and Use Self-Efficacy (MUSE) Scale. It measures patients' self-efficacy in understanding and using medication.
Barriers to adherence and problems with adherence behavior | Up to 6 months post-baseline
  Will be assessed by the Adherence Starts With Knowledge 12 Questionnaire (ASK-12).
Beliefs in medications | Up to 6 months post-baseline
  Will be measured using the Beliefs in Medicines Questionnaire (BMQ).
Individual illness perceptions | Up to 6 months post-baseline
  Will be assessed using Brief-Illness Perceptions Questionnaire (B-IPQ) that includes survey items assessing individual illness perceptions along the cognitive domains of the self-regulatory model as well as emotional responses to having CML.
Self-efficacy for medication use | Up to 6 months post-baseline
  Will be measured using the 13-item Self-efficacy for Appropriate Medication Use Scale (SEAMS).
Health-related quality of life (HRQoL) | Up to 6 months post-baseline
  Will be assessed using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) Questionnaire consisting of leukemia-specific sub scale.
Health-related quality of life (HRQoL) | Up to 6 months post-baseline
  Will be assessed using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) Questionnaire consisting of a set of general HRQoL questions (Functional Assessment of Cancer Therapy-General [FACT-G])
Self-efficacy for managing symptoms | Up to 6 months post-baseline
  Will be measured by a modified version of Lorig's Chronic Disease Self-Efficacy Scale for managing symptoms.
Affect | Up to 6 months post-baseline
  The Intrusion subscale of the Revised Impact of Events Scale (RIES) will be used to assess affective distress concerning TKI.
Social Support | Up to 6 months post-baseline
  Will be measured using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS assesses perceptions of support received from family, friends, and significant others.
Usefulness and satisfaction of txt4TKI | Up to 6 months post-baseline
  Patient interviews will explore key domains including perceived usefulness, how well txt4TKI address their concerns, whether there are additional issues they would like to see included and the characteristics of the text messaging (TXT). Client Satisfaction Questionnaire (CSQ-8) structured measures will ask participants to rate the usefulness and satisfaction of txt4TKI and how likely they would recommend the program to others.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States